CLINICAL TRIAL: NCT07407231
Title: Efficacy Of Combination Chemotherapy And Ablative Radiotherapy (SBRT) In The First-Line Treatment Of Locally Advanced Inoperable Pancreatic Cancer
Brief Title: Combined Chemotherapy And Ablative Radiotherapy (SBRT) As First-Line Treatment In Locally Advanced Inoperable Pancreatic Cancer (SBRT-PANC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OI-LJ-PANC-SBRT-2021; ARRS-13541 (Other: Onkološki Inštitut Ljubljana)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: SBRT; Stereotactic Body Radiotherapy

STUDY DESIGN:
Intervention Model Description: Participants receive standard first-line chemotherapy followed by ablative stereotactic body radiotherapy (SBRT) in the absence of progression, with continuation of systemic therapy according to clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Chemotherapy Followed by Ablative SBRT (Experimental): Participants receive standard first-line systemic chemotherapy. Patients without disease progression after initial chemotherapy undergo ablative stereotactic body radiotherapy (SBRT) to the primary pancreatic tumor, followed by continuation of systemic therapy according to institutional practice.
  Interventions: Radiation: Ablative Stereotactic Body Radiotherapy (SBRT); Drug: Standard First-Line Chemotherapy

INTERVENTIONS:
Radiation: Ablative Stereotactic Body Radiotherapy (SBRT) — Ablative stereotactic body radiotherapy (SBRT) delivered to the primary pancreatic tumor after initial chemotherapy in patients without disease progression.
Drug: Standard First-Line Chemotherapy — Standard first-line systemic chemotherapy administered according to institutional guidelines (e.g., modified FOLFIRINOX or gemcitabine plus nab-paclitaxel), followed by continuation of systemic therapy after SBRT as clinically indicated.

SUMMARY:
This prospective interventional clinical study evaluates the efficacy and safety of combining systemic chemotherapy followed by ablative stereotactic body radiotherapy (SBRT) as first-line treatment in adult patients with locally advanced, inoperable pancreatic cancer.

The study aims to determine the response rate after SBRT delivered following initial chemotherapy, as well as time to disease progression and treatment-related toxicity. Patients receive standard first-line chemotherapy and, in the absence of disease progression, undergo ablative SBRT to the primary tumor, followed by continuation of systemic therapy according to clinical practice.

The study is conducted in Slovenia, with patient enrollment expanded to additional participating clinical centers following an approved amendment.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly aggressive malignancy with poor prognosis. In patients with locally advanced pancreatic cancer (LAPC) who are not candidates for surgical resection, systemic chemotherapy is the standard first-line approach. However, local tumor progression remains a major cause of morbidity and mortality. Stereotactic body radiotherapy (SBRT) enables delivery of high-dose ablative radiation to the primary tumor while minimizing exposure of surrounding organs at risk.

This prospective interventional study investigates a combined treatment strategy consisting of initial systemic chemotherapy followed by ablative SBRT in adult patients with locally advanced, inoperable pancreatic cancer.

Eligible patients receive first-line systemic chemotherapy according to standard clinical practice. Patients without progression after initial chemotherapy are treated with ablative SBRT directed to the primary pancreatic tumor. After completion of SBRT, patients may continue systemic treatment based on clinical evaluation and institutional practice.

The primary objective of the study is to evaluate the response rate following ablative SBRT after initial chemotherapy. Secondary objectives include evaluation of time to disease progression and safety/tolerability of the combined treatment approach, including acute and late treatment-related toxicity.

The study is conducted as a non-randomized prospective clinical trial. Following an approved amendment, additional clinical centers in Slovenia were included to support recruitment and increase the number of enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years and older

Locally advanced, inoperable pancreatic cancer

Treated with first-line systemic chemotherapy followed by stereotactic body radiotherapy (SBRT) at participating centers

Ability to provide written informed consent

Exclusion Criteria:

Metastatic pancreatic cancer

Prior systemic therapy for locally advanced pancreatic cancer (one or more previous lines of systemic treatment)

Disease progression after initial chemotherapy prior to SBRT

Any condition that, in the investigator's opinion, would interfere with study participation or evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Response Rate After SBRT | Up to 12 weeks after completion of SBRT
  Proportion of participants achieving treatment response after initial chemotherapy followed by ablative stereotactic body radiotherapy (SBRT), assessed by radiologic imaging (CT/MRI) according to standard response evaluation criteria.

SECONDARY OUTCOMES:
Time to Disease Progression | Up to 36 months
  Time from start of first-line chemotherapy to radiologic or clinical disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No